CLINICAL TRIAL: NCT05387655
Title: Long Term Assessment of Infectious Diseases and Immune Mediated Disorders After BCG (re)Vaccination
Brief Title: Long Term Effects of BCG Vaccination on Infectious and Immune Mediated Diseases
Acronym: BCG-LT
Status: Active, not recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: UMC Utrecht (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-13462
Record Dates: First submitted 2022-05-12; First posted 2022-05-24 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: BCG Vaccination Reaction; Infections; Inflammation; COVID-19
MeSH Terms: conditions — Infections; Inflammation; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- BCG vaccination: People who received a BCG vaccination in the prior BCG-CORONA-ELDERLY or BCG-PRIME study
  Interventions: Biological: BCG
- Placebo vaccination: People who received a placebo vaccination in the prior BCG-CORONA-ELDERLY or BCG-PRIME study
  Interventions: Biological: Placebo vaccine

INTERVENTIONS:
Biological: BCG — BCG vaccination
  Groups: BCG vaccination
Biological: Placebo vaccine — Placebo vaccination
  Groups: Placebo vaccination

SUMMARY:
Rationale: The effects of BCG vaccination have been only sporadically studied in the elderly, and the long-term effects of the vaccination have not been studied until now. There is evidence that BCG vaccination beneficially influences susceptibility and severity of infectious and inflammatory diseases; however, the specifics, extent and duration of these effects are not known yet. With this observational study we would like to determine the extent of these effects in the elderly.

Objective: To identify any long term effects of BCG vaccination on the incidence of infectious and inflammatory diseases may have in the elderly

Study design: Cohort study with a duration of 5 years

Study population: Older adults who participated in two large randomized BCG vaccination trials in 2020/2021 (BCG-CORONA-OUDEREN, BCG-PRIME), who have consented to be contacted for further studies

Main study parameters/endpoints:

The incidence of infectious and inflammatory diseases in the placebo- vs. BCG-vaccinated individuals

ELIGIBILITY:
Inclusion Criteria:

* Completed participation in the BCG-CORONA-ELDERLY or BCG-PRIME study
* Given consent to be approached for further studies

Exclusion Criteria:

* Has received a BCG vaccination after the BCG-CORONA-ELDERLY or BCG-PRIME study

Inclusion Criteria from BCG-PRIME:

* Age ≥60 years
* Meeting at least one of the following criteria:

  1. Having a chronic somatic disease*
  2. Having undergone major surgery**
  3. Planned to be discharged from the hospital or discharged from the hospital less than 6 weeks ago; a hospital admission is defined as an overnight stay. Departments of interest are those that in the opinion of the principle investigator admit mostly vulnerable elderly and include but are not limited to: cardiology, pulmonology, internal medicine, neurology.
  4. Attending the thrombosis care service * Chronic somatic diseases do not include risk factors such as hypertension or obesity unless the participant receives medication targeted against the risk factor.

     * Major surgery is any invasive operative procedure in which a more extensive resection is performed, e.g. a body cavity is entered, organs are removed, or normal anatomy is altered. In general, if a mesenchymal barrier is opened (pleural cavity, peritoneum, meninges), the surgery is considered major

Exclusion criteria from BCG-PRIME:

* Fever (>38 ºC) within the past 24 hours
* Suspicion of current active viral or bacterial infection; the requirement to finish an antibiotic course upon discharge is not an exclusion criterion when the infection is controlled in the opinion of the attending physician
* Vaccination with live vaccine in the past four weeks or planned vaccination with live vaccine during the next four weeks
* Severely immunocompromised participants. This exclusion category comprises:

  1. known infection by the human immunodeficiency virus (HIV-1);
  2. neutropenic with less than 500 neutrophils/mm3;
  3. solid organ transplantation;
  4. bone marrow transplantation;
  5. hematological malignancy;
  6. chemo-, radio- or immunotherapy for solid organ malignancy in the past 6 months;
  7. primary immunodeficiency;
  8. severe lymphopenia with less than 400 lymphocytes/mm3;
  9. treatment with any immunosuppressant drugs such as anti-cytokine therapies, and treatment with oral or intravenous steroids defined as daily doses of >10 mg/day or a cumulative dose of >700 mg prednisone or equivalent for other corticosteroids in the three months prior to enrolment, or probable use of oral or intravenous steroids in the following four weeks;
  10. receiving chronic renal replacement therapy.
* Known history of a positive Mantoux or active TB; prior BCG vaccination or a positive Mantoux test after BCG vaccination without confirmation of TB are NOT an exclusion criterion.
* Born in a country with high incidence of TB (see supplement B)
* Active participation in another research study that involves BCG administration
* History of documented COVID-19 (self-reported by the participant: either confirmed by a microbiological test or with clinical diagnosis during hospitalization)
* Not able to perform the study procedures as judged by the attending physician
* Legally incapacitated or unwilling to provide informed consent

Inclusion criteria from BCG-CORONA-ELDERLY:

* Adult (≥ 60 years)
* Written informed consent

Exclusion criteria from BCG-CORONA-ELDERLY:

* Fever (>38 ºC) within the past 24 hours
* Suspicion of current active viral or bacterial infection
* Expected vaccination during the first three months of the study period
* Severely immunocompromised subjects. This exclusion category comprises: a) subjects with known infection by the human immunodeficiency virus (HIV-1); b) neutropenic subjects with less than 500 neutrophils/mm3; c) subjects with solid organ transplantation; d) subjects with bone marrow transplantation; e) subjects under chemotherapy; f) subjects with primary immunodeficiency; g) severe lymphopenia with less than 400 lymphocytes/mm3; h) treatment with any immunosuppressant drugs such as anti-cytokine therapies, and treatment with oral or intravenous steroids defined as daily doses of 10mg prednisone or equivalent for longer than 3 months, or probable use of oral or intravenous steroids in the following four weeks
* Active solid or non-solid malignancy or lymphoma within the prior two years
* Active participation in another research study that involves BCG administration

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of participants who previsouly participated in the BCG-CORONA-ELDERLY or BCG-PRIME study and gave consent for further participation. All former participants will receive an invitation to join this LongTerm study.
Sampling Method: Non-Probability Sample
Enrollment: 4292 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of infectious and inflammatory disease | One year after the end of participation in the BCG-CORONA-ELDERLY or BCG-PRIME study; the questions in the questionnaire are about events 'in the last year' (so from the moment of sending the questionnaire)

SECONDARY OUTCOMES:
Incidence of various non-communicable diseases | One year after the end of participation in the BCG-CORONA-ELDERLY or BCG-PRIME study; the questions in the questionnaire are about events 'in the last year' (so from the moment of sending the questionnaire)

OTHER OUTCOMES:
Use of antibiotics | One year after the end of participation in the BCG-CORONA-ELDERLY or BCG-PRIME study; the questions in the questionnaire are about events 'in the last year' (so from the moment of sending the questionnaire)
Vaccination status | One year after the end of participation in the BCG-CORONA-ELDERLY or BCG-PRIME study; the questions in the questionnaire are about events 'in the last year' (so from the moment of sending the questionnaire)
Incidence of infectious and inflammatory diseases | One year since last questionnaire (so between 1-2 years after completion of original BCG trial)
Incidence of infectious and inflammatory diseases | One year since last questionnaire (so between 2-3 years after completion of original BCG trial)
Incidence of infectious and inflammatory diseases | One year since last questionnaire (so between 3-4 years after completion of original BCG trial)
Incidence of infectious and inflammatory diseases | One year since last questionnaire (so between 4-5 years after completion of original BCG trial)
Incidence of various non-communicable diseases | One year since last questionnaire (so between 1-2 years after completion of original BCG trial)
Incidence of various non-communicable diseases | One year since last questionnaire (so between 2-3 years after completion of original BCG trial)
Incidence of various non-communicable diseases | One year since last questionnaire (so between 3-4 years after completion of original BCG trial)
Incidence of various non-communicable diseases | One year since last questionnaire (so between 4-5 years after completion of original BCG trial)
Use of antibiotics | One year since last questionnaire (so between 1-2 years after completion of original BCG trial)
Use of antibiotics | One year since last questionnaire (so between 2-3 years after completion of original BCG trial)
Use of antibiotics | One year since last questionnaire (so between 3-4 years after completion of original BCG trial)
Use of antibiotics | One year since last questionnaire (so between 4-5 years after completion of original BCG trial)
Vaccination status | One year since last questionnaire (so between 1-2 years after completion of original BCG trial)
Vaccination status | One year since last questionnaire (so between 2-3 years after completion of original BCG trial)
Vaccination status | One year since last questionnaire (so between 3-4 years after completion of original BCG trial)
Vaccination status | One year since last questionnaire (so between 4-5 years after completion of original BCG trial)

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No